CLINICAL TRIAL: NCT02302417
Title: The Utility of a Clinical Questionnaire to Identify Subjects With Features of Both Asthma and COPD
Brief Title: Study Assessing Utility of a Clinical Questionnaire to Identify Subjects With Features of Both Asthma and Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201703
Record Dates: First submitted 2014-11-06; First posted 2014-11-27 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Asthma; Asthma-COPD Overlap Syndrome; Clinical Questionnaire; COPD; ACOS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Other): Approximately 1000 subjects with clinical diagnoses of asthma and/or COPD or clinical presentations suggestive of either or both will be included. Subjects will undergo spirometry assessments and also will be asked a series of questions by a qualified health care practitioner using a questionnaire containing 41 questions concerning their respiratory condition.
  Interventions: Procedure: Spirometry; Other: ACOS clinical questionnaire

INTERVENTIONS:
Procedure: Spirometry — Classification of respiratory diseases by Spirometry will be performed to differentiate subjects between Asthma only, ACOS, and COPD only. Spirometry obtained from measurements in the past 6 months is acceptable for purposes of this study. For subjects without spirometry in the past 6 months, spirometry will be performed to obtain pre- and post-bronchodilator Forced Expiratory Volume in one second (FEV1), Forced Vital Capacity (FVC) and reversibility
Other: ACOS clinical questionnaire — The 41-question questionnaire includes questions concerning the following: a) response to bronchodilator, b) disease progression, c) variations in symptom, d) atopic history, e) symptom triggers, f) vagal bias, g) burden of disease, h) symptom presentation, i) emotional aspects, and j) age of onset. In addition, two questions will capture patient perception of his/her respiratory disease and the physician's diagnosis

SUMMARY:
The primary objective of the study is to identify demographic and non-spirometric clinical features predictive of the asthma-COPD overlap population. The study aims to explore and identify characteristics of the Asthma-COPD Overlap Syndrome (ACOS) patient's clinical profile that enable clinical differentiation from subjects with a primary diagnosis of either asthma alone (without persistent obstruction) or COPD alone (without reversibility). The study is designed as a targeted medical history survey which consists of a 41-item questionnaire, which will be administered by a qualified health care practitioner at the time a subject's medical history is taken. The questionnaire has been developed to elicit specific details of the respiratory history, including the following: bronchodilator use, disease progression, variation in symptoms, atopic history, symptom triggers, vagal bias, burden of disease, symptom presentation, co morbidities and age of onset. In addition, demographic information, standard medical history, co morbidity and spirometric results will also be obtained and analyzed in conjunction with the questionnaire results. Approximately 1000 subjects are required for the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* Subject has been diagnosed as having asthma and/or COPD.
* Informed consent is required for independent sites initiating this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1215 (Actual)
Dates: Start 2015-01-01; Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-28 (Actual)

PRIMARY OUTCOMES:
Summary of spirometry data: forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) | Day 1
  FEV1 measures how much air a person can exhale during a forced breath in 1 second. FVC is the total amount of air exhaled during the FEV test. FEV1 and FVC were performed on Day 1 (pre- and post-bronchodilator) using spirometry. Spirometry results obtained within 6 months and were used for this study. For participants without spirometry in the past 6 months, spirometry was performed to obtain pre- and post-bronchodilator FEV1, FVC.
Summary of spirometry data: Reversibility | Day 1
  Questionnaire designed to clinically differentiate participants with ACOS from patients who have either asthma alone (i.e. without persistent obstruction) or COPD alone (i.e., non-reversible). Spirometry results obtained within 6 months and were used for this study. For participants without spirometry in the past 6 months, spirometry was performed to obtain pre- and post-bronchodilator FEV1, FVC and reversibility.
Number of participants with response to Bronchodilators (Questionnaire Items 1 and 2) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Response to bronchodilators was one domain in which, participants had to answer questions (Q)1-2 (Q1: How well does your participant's quick relief inhaler (rescue inhaler) provide symptom relief? and Q2: How often does the participant need to keep a rescue inhaler with him/her?) regarding rescue inhaler and need to keep inhaler with participants Responses were recorded as No relief, Relief and No need, Need. Number of participants with such responses were recorded.
Number of participants with disease progression (Questionnaire Item 3) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Disease progression was one domain in which, participants had to answer question (Q3: How does the participant describe his/her respiratory disease over the past two (2) years?) regarding disease progression over the past two years with responses like: getting worse or same/some better/some worse. Number of participants with such responses were recorded.
Number of participants with Variation in symptoms (Questionnaire Items 4-10) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Variation in symptoms was one domain in which, participants had to answer questions 4 to 10 which included questions regarding respiratory symptoms, night-time awakenings due to symptoms, respiratory symptoms during day and night, good/bad days regard to breathing, good and bad days difference, how quickly a good day changes to bad, how long until the bad respiratory symptoms return to normal. Number of participants with such responses were reported.
Number of participants with atopic history (Questionnaire Items 11 and 12) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Atopic history was one domain in which, participants had to answer questions 11 and 12 (Q11: Has the participant ever had nasal allergies or eczema? and Q12: How many members of the participant's immediate biological family have had asthma, nasal allergies, or eczema? )which included questions regarding nasal allergies or eczema and how many members of the participant's immediate biological family had asthma, nasal allergies, or eczema. Number of participants with responses to these questions were reported.
Number of participants with atopic history (Questionnaire Items 13-15) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Atopic history was one domain in which, participants had to answer questions 13-15 (Q13: Do the subject's respiratory symptoms get worse after exposure to pollen or pets?, Q14: Do the subject's respiratory symptoms get worse after exposure to cold air or weather changes?, Q15: Do the subject's respiratory symptoms get worse with exposure to air pollution or noxious fumes? ). Responses of participants as yes or no were recorded for these questions.
Number of participants with vagal bias (Questionnaire Items 16 and 17) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. vagal bias was one domain in which, participants had to answer questions 16 and 17 (Q16: Does the participant react emotionally to distress (e.g., cry easily during a sad film)?, Q17: How much of an impact does emotional distress have on the participant's respiratory symptoms? ). Number of participants with response to these questions were reported.
Number of participants with burden of disease (Questionnaire Items 18-24) | Day 1
  ACOS Medical history questionnaire is a disease specific questionnaire to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Burden of disease was a domain in which, participants had to answer questions 18-24 (Q18: If the participant stops taking his/her regular respiratory medications, how do his/her respiratory symptoms change?, Q19: How many days in a week does the participant typically have respiratory symptoms during the day?, Q20: How often does the participant typically have respiratory symptoms at night?, Q21: On average how frequently does the participant use rescue medication?, Q22: How often do the participant's respiratory symptoms disturb their sleep?, Q23: How much impact do the participant's respiratory symptoms have on their energy level?, Q24: How often would the participant describe themselves as feeling anxious?). Number of participants with response to these questions were reported.
Number of participants with symptom presentation (Questionnaire Items 25-34) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Burden of disease was one domain in which, participants had to answer questions 25-34 which included questions regarding presentation of symptoms like cough, breathlessness, sputum production. Responses to these questions were recorded. Question 33 was a 5 part question with cough, breathlessness, sputum production as the most bothersome symptom (MBS) Number of participants with responses to the questions were reported.
Number of participants with emotional response by Sex (Questionnaire Items 35 and 36) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Emotional Response was one domain in which, participants had to answer questions 35-36 (Q35: How often would the participant describe themselves as feeling depressed?, Q36: How scared or worried is the participant about his/her lung function?)for males and females was collected and number of participants with responses were reported.
Summary of age of onset (Questionnaire Items 37 and 38) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Age of onset was one domain in which, participants had to answer questions 37 and 38 (Q37: How old was the participant when he/she first used an inhaler (for asthma or COPD)?, Q38: How old was the participant when he/she first used an inhaled corticosteroid on a regular basis for his/her respiratory condition (asthma or COPD)?). Least square mean was presented.
Number of participants with perception of respiratory disease (Questionnaire Items 39-40) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. Patient Perception of respiratory disease was one domain in which, participants had to answer questions 39-40 (Q39: Does the participants consider themselves to have asthma, COPD or both?, Q40: Does this participants have asthma, COPD or both?). Number of participants with both responses were collected and presented.
Number of participants with clinical features most helpful in diagnosis (Questionnaire Item 41) | Day 1
  ACOS Medical history questionnaire is a disease specific (asthma and/or COPD) questionnaire administered by a qualified health care practitioner to assess the clinical features of asthma and/or COPD. Items were grouped in 10 different domains. clinical features most helpful in diagnosis was one domain in which, participants had to answer question item 41 which was regarding various clinical features like age of onset, symptom presentation, variation in symptoms, timing of symptoms, symptom persistence, previous environmental exposure, tobacco smoking history, airflow limitation variability, lung function measures, nature of disease, previous doctor diagnosis, family history, response to short-acting bronchodilator, response to inhaled corticosteroid (ICS), chest x-ray findings, symptom triggers. Number of participants with responses to these questions were reported.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (12):
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (7):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Germany (6):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Berlin
- Russia (5):
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
- Ukraine (3):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv